CLINICAL TRIAL: NCT02415517
Title: Cognitive Training in Heart Failure Study (CogTrain-HF)
Acronym: CogTrain-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Collaborators: Deutsche Stiftung für Herzforschung (Other)
Responsible Party: Principal Investigator, Sonja Wedegärtner, Dipl. Psych., Universität des Saarlandes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CogTrain-HF
Record Dates: First submitted 2015-04-02; First posted 2015-04-14 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Congestive Heart Failure; Cognitive Impairment
Keywords: Cognitive training; Cognitive impairment; Heart failure; Cognition
MeSH Terms: conditions — Heart Failure; Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Pre-Test, Intervention, Post-Test, Follow-Up
Who Masked: Participant
Masking Description: Participants were enrolled in Treatment-Group, Waitinglist-Group, or Shamtraining-Group
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental group (Experimental): Intervention: Cognitive Training
  Interventions: Behavioral: Cognitive training
- Active control group (Active Comparator): Intervention: Test of general knowledge
  Interventions: Behavioral: Test of general knowledge
- Passive control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Cognitive training — Cognitive training on computer. Six sessions with different tasks: "Tiere merken" & "Räumlich visuelles Training" (application BrainTwister) and "Taskswitching" (programmed with eprime)
  Arms: Experimental group
Behavioral: Test of general knowledge — Training of general knowledge on computer. Six sessions with different topics.
  Arms: Active control group

SUMMARY:
The daily routine in clinical settings often showed cognitive impairments in patients with congestive heart failure, particularly in terms of executive functions, episodic memory, perceptual speed and attention. It is assumed that cognitive impairments in patients with congestive heart failure may lead to deficits in medication-adherence and self-care abilities, resulting in increased healthcare costs. Recent studies reported performance improvements after cognitive training that transferred to new, untrained tasks and abilities in healthy subjects across a wide range of ages. This study investigates the effects of cognitive training in patients with congestive heart failure.

DETAILED DESCRIPTION:
Cognitive functions of patients with congestive heart failure (NYHA II-III) before (pretest) and after (posttest) cognitive-training intervention are investigated. Changes in cognitive functions are compared to changes in two control groups: 1) age and gender matched active control group 2) age and gender matched passive waiting list control group.

The neuropsychological test battery applied at pretest and posttest includes measures of episodic memory, working memory, short-term memory, executive functions, perceptual speed and intelligence. In addition, the investigators apply standardized questionnaires of self-assessed quality of life, cognitive functioning in daily life, selfcare, and psychological well-being (depression, anxiety and personality). Relevant physiological data such as ejection fraction, heartrate, N-terminal pro brain natriuretic peptide (NT-pro-BNP) as well as drug blood level are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Congestive heart failure
* NYHA II-III

Exclusion Criteria:

* Psychosis
* Dementia
* Major depression
* Reanimation (<3month)
* Patients with assist device system

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-01; Primary Completion 2019-06-03 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Training effects | 3 weeks
  Improvement in performance in the last trainingssession compared with the performance in the first trainingssession. Performance will be assessed by computesoftware.

SECONDARY OUTCOMES:
Transfer effects | 5 weeks
  Transfer effects are measured by comparing cognitive functions in patients with congestive heart failure before and after cognitive training. Cognitive functions will be assessed by different paper-and-pencil tests and computerbased tests.
Changes in quality of life and psychological well-being | 5 weeks
  Changes in quality of life and psychological well-being as the result of cognitive training measured by psychological questionnaires and tests.
Long-term benefits of cognitive training in patients with congestive heart failure. | 6 month
  Follow-up assessment by 6 months after training. Long-term benefits will be measured by different paper-and-pencil tests and computerbased tests as well as psychological questionnaires and tests.
Compliance with medication | 5 weeks
  Compliance with medication measured as serum level of medication and heart failure-specific self-care duties.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Kindermann, PD Dr.med., Study Director — University Hospital, Saarland; Julia Karbach, Prof., Study Director — Goethe-Universität Frankfurt am Main; Sonja Wedegärtner, Dipl.Psych., Principal Investigator — University Hospital, Saarland; Maxie Bunz, Dipl.Psych., Principal Investigator — University Hospital, Saarland; Michael Böhm, Prof., Study Chair — University Hospital, Saarland
Locations (2):
- Germany (2):
  - Department of Educational Science, Saarland University, Frankfurt am Main, Hesse
  - Clinic for Internal Medicine, Cardioloy, Angioloy, and Internal Intensive Care Medicine, Saarland University Hospital, Homburg, Saarland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Wedegartner SM, Schwantke I, Kindermann I, Karbach J. Predictors of heart-focused anxiety in patients with stable heart failure. J Affect Disord. 2020 Nov 1;276:380-387. doi: 10.1016/j.jad.2020.06.065. Epub 2020 Jul 15. PMID 32871668